CLINICAL TRIAL: NCT01043367
Title: Efficacy of Deprexil Administration in Subjects With Signs and Symptoms of Depression.
Brief Title: Deprexil in Subjects With Signs and Symptoms of Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Maria de la Concepción Valdivia Alarcón, "Heroes del Moncada" Polyclinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0908-CU
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Depression
Keywords: Depression; Dietary supplement; Deprexil
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Deprexil
  Interventions: Dietary Supplement: Deprexil
- B (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Deprexil — One 600 mg Deprexil tablet (Orally administered) half an hour after each meal (breakfast, lunch and dinner), for 24 weeks. A 20 minutes relaxation psychotherapy will also be provided once a week.
  Arms: A
Dietary Supplement: Placebo — One Placebo tablet (Orally administered) half an hour after each meal (breakfast, lunch and dinner), for 24 weeks. A 20 minutes relaxation psychotherapy will also be provided once a week.
  Arms: B

SUMMARY:
The purpose of the study is to assess the efficacy of DEPREXIL administration in combination with relaxation psychotherapy in the treatment of patients with signs and symptoms of depression. The duration of this double-blind placebo controlled phase 3 clinical trial will be 24 weeks. The estimated number of persons to be recruited and randomized for the study is 200.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate symptoms and signs of depression for more than 3 months and less than 3 years of duration.
* Signed informed consent

Exclusion Criteria:

* Severe symptoms and signs of depression or Suicide proneness.
* Pregnancy or breastfeeding
* Receiving other experimental drug
* Use of anti-depressive medication within 15 days

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Functional capabilities at week 24 (end of the treatment) | 24 weeks
Social capabilities at week 24 (end of the treatment) | 24 weeks
Psycho-affective capabilities at week 24 (end of the treatment) | 24 weeks
Behavioral capabilities at week 24 (end of the treatment) | 24 weeks

SECONDARY OUTCOMES:
Tolerability to Deprexil at week 24 (end of the treatment) | 24 weeks
Symptoms of depression at week 24 (end of the treatment) | 24 weeks
Signs of depression at week 24 (end of the treatment) | 24 weeks
Clinical symptoms of baseline disease at 24 weeks (end of the treatment) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria de la Concepción Valdivia Alarcón, MD, Principal Investigator — "Heroes del Moncada" Polyclinic
Locations (1):
- "Heroes del Moncada" Polyclinic, Havana, La Habana, Cuba